CLINICAL TRIAL: NCT04679974
Title: Melodic-based Communication Therapy for Promoting Spoken Language Development in Individuals With Nonverbal Autism Ages: 3:0 - 10:11
Brief Title: Melodic-based Communication Therapy for Promoting Spoken Language Development in Individuals With Nonverbal Autism
Acronym: MBCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Karen Mainess, Assistant Professor, Loma Linda University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5170235
Record Dates: First submitted 2020-12-17; First posted 2020-12-22 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Nonverbal and Low Verbal Autism
Keywords: MBCT; Nonverbal autism; low verbal autism

STUDY DESIGN:
Intervention Model Description: ABA design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MBCT treatment (Experimental): Melodic-based communication treatment
  Interventions: Behavioral: Melodic-based Communication Therapy

INTERVENTIONS:
Behavioral: Melodic-based Communication Therapy — General procedures involved in (M.B.C.T.) are as follows: 25 common first words are selected as the targets (e.g., apple, ball, car, dog, cat, eat, go, etc.). Pictures and objects will be used as stimulus items. The top 3-5 incentives as identified by parent survey will be given according to the therapies specific reinforcement schedule. All treatment and evaluation sessions will be videotaped for future/further analysis and verification purposes. For the purposes of the study design, the same 25 words will be used for all participants.
  Participants will first listen to the target word set to a melodic tone and rhythm on a compact disc (CD). Clinicians will present the stimulus item (e.g., apple) prior to beginning the steps. Therapy will then progress from clapping and singing the melody to answering sung questions and finally to answering spoken questions with the target word

SUMMARY:
The purpose of this study is to determine the efficacy of Melodic Based Communication Therapy (M.B.C.T.) for increasing oral expressive skills in nonverbal children with autism spectrum disorders. MBCT has previously been shown to facilitate an improvement in expressive vocabulary, verbal imitative abilities, number of vocalizations, and social language development in nonverbal children with autism ages 5-7. However, earlier studies were small and did not examine the effects of M.B.C.T. on a younger and older population. This study will examine its effectiveness across a broader sample group. Additionally, this study will examine further predictors of success including but not limited to chronological age, developmental age, the frequency of repetitive/stereotypic behaviors, receptive language score, and social language score.

DETAILED DESCRIPTION:
The study will be a repeated measures design as assessments will be taken at baseline and on a weekly basis (baseline, weeks 1-4). All participants in the study will receive Melodic Based Communication Therapy (M.B.C.T.). General procedures involved in (M.B.C.T.) are as follows: 25 common first words are selected as the targets (e.g., apple, ball, car, dog, cat, eat, go, etc.). Pictures and objects will be used as stimulus items. The top 3-5 incentives as identified by parent survey will be given according to the therapies specific reinforcement schedule. All treatment and evaluation sessions will be videotaped for future/further analysis and verification purposes. For the purposes of the study design, the same 25 words will be used for all participants.

4. Subjects will be male and female children diagnosed with autism.

5. Subjects will be between 3 years 0 months and 10 years 11 months of age.

6. In total, subject participation will last approximately 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male and female children with autism ages 3-years-0-months to 10-years-11-month who meet the criterion for nonverbal (defined as less than 10 words ever spoken expressively and no functional verbal communication)

Exclusion Criteria:

* Individuals receiving other language or articulation treatments or therapy at the time of the study, unable to regularly attend four 30 min sessions of therapy weekly for 4 weeks, a history of severe hearing impairment, severe visual impairment/ blindness, a diagnosis of an organic impairment of oral or laryngeal structures, or a signiﬁcant medical illness or condition which would prevent the child's participation in the treatment procedures. These conditions include, but are not limited to cerebral palsy, paraplegia, spina biﬁda, uncontrolled seizures, dysarthria, and amputation of arm(s).

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2018-06-17 (Actual); Primary Completion 2018-08-16 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Number of spoken words | 4 weeks
  Pre/post measures include: number of words reported in home environment by parent pre-vs. post, CASL-2 Pragmatic Language raw score pre-vs. post, number of imitative attempts pre-vs. post, number of words correct in response to the question, "what is this?" and number of vocalizations in response to the question, "what is this?"
Frequency of repetitive and stereotypical behaviors | 4 weeks
  Frequency of repetitive or stereotypic movements will be analyzed in the first week of treatment (stimming behavior). This will be evaluated as follows: onset/offset and duration of the behaviors to determine frequency. This will be evaluated by an independent observer through video analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Loma Linda University, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No